CLINICAL TRIAL: NCT01668550
Title: A Cancer Research UK Phase I Study to Determine the Maximum Tolerated Dose of the Oral Src/Abl Inhibitor AZD0424, and to Identify Tolerable and Effective AZD0424 Combination Regimens for the Treatment of Advanced Solid Tumours
Brief Title: A Phase I Study of AZD0424 Alone and in Combination in Advanced Solid Tumours
Acronym: AZD0424
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Single agent phase completed, insufficient supportive preclinical data to proceed with combination phase
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/07/061
Record Dates: First submitted 2012-05-31; First posted 2012-08-20 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2016-07

CONDITIONS: Advanced Solid Tumours
Keywords: Phase I; Src/Abl inhibitor; Solid Tumours; Cancer
MeSH Terms: conditions — Neoplasms | interventions — AZD-0424

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD0424 — AZD0424 will be administered as a flat dose orally once a day. One treatment cycle consists of 28 days of continuous drug administration with AZD0424, with the flexibility to introduce treatment breaks if required due to cumulative toxicity.
  Combination agents and treatment regimen with AZD0424 will be confirmed and approved at a later date.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of the oral Src/Abl inhibitor AZD0424, and to find tolerable and effective AZD0424 combination regimens for the treatment of advanced solid tumours

DETAILED DESCRIPTION:
AZD0424 is a potent orally available, potent (IC50 approximately 4 nM) inhibitor of Src and ABL1 kinases with additional activity against Src family kinase (SFK) members including Yes and Lck. AZD0424 was selective for SFKs and ABL1 kinase over C-terminal Src kinase (a negative regulator of Src) and a range of other kinase targets. The anti-cancer activity of AZD0424 is thought to be mediated primarily by anti-migratory and anti-invasive signalling and, as such, it is expected that in the late stage cancer setting strong signals of efficacy with this compound used as a single agent are unlikely, requiring it to be administered in combination with other anti-cancer agents.

In summary the study will be performed in four main stages:

* AZD0424 monotherapy, dose escalation: Phase Ia single agent (AZD0424) dose escalation study to determine the MTD.
* AZD0424 monotherapy, dose expansion: Phase Ib single agent dose expansion at MTD (up to six additional patients may be recruited in order to provide paired tumour biopsies for PD analysis).
* Combination arm dose escalation: Provided that it is deemed appropriate (after review of available clinical data from the monotherapy part of the trial, and available preclinical and published data on the combination), a Phase Ia dose escalation arm of AZD0424 in combination with the selected agent will proceed to determine the MTD for the combination and a recommended Phase II dose.
* Combination arm dose expansion: Phase Ib combination arm using the recommended Phase II dose for both AZD0424 and the combination agent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven solid tumour, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient or for whom there is the prospect of clinical benefit
* Life expectancy of at least 12 weeks
* World Health Organisation (WHO) performance status of 0-2
* Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) before the patient receives AZD0424

  * Haemoglobin (Hb) ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x (ULN) Either: Calculated creatinine clearance ≥ 50 mL/min Or Or Isotope Clearance measurement ≥ 50 mL/min (uncorrected)
* 18 years or over
* Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up
* MTD Expansion cohorts only: A tumour which is safely accessible for biopsy (single and combination)

Exclusion Criteria:

* Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C and four weeks for investigational medicinal products) before treatment.
* Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the DDO should not exclude the patient.
* Symptomatic brain metastases (if brain metastases are present they must have been stable for > 3 months).
* Patients with evidence of interstitial lung disease (bilateral, diffuse, parenchymal lung disease).
* Patients with a peanut allergy will be excluded.
* Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrollment and agree to use two highly effective forms of contraception as detailed in the protocol are considered eligible.
* Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception as detailed in the protocol). Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
* Major thoracic or abdominal surgery from which the patient has not yet recovered.
* At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
* Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
* Resting ECG with measurable QTc interval of >480 msec (mean value and manually verified) of at least 3 time points within a 24 hour period.
* Concurrent hypotension defined as a baseline supine blood pressure (BP) systolic < 90 mmHg.
* Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA]), prior history of cardiac ischaemia or prior history of cardiac arrhythmia within 6 months. Coronary angioplasty or stenting in the previous 12 months.
* Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase Ia/Ib study of AZD0424 single agent and in combination. Participation in an observational, counseling or psychological trial would be acceptable.
* Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Establishing the Maximum Tolerated Dose (MTD) of AZD0424 alone and in combination
Determining the causality and duration of adverse events observed during the study according to NCI CTCAE Version 4.02

SECONDARY OUTCOMES:
Determining the correlation between PK studies and toxicity and/or efficacy.
Measurement of urinary and serum N terminal Telopeptide (NTx) and serum C-terminal peptide (CTx) levels before the first AZD0424 administration and then following first AZD0424 administration, to evaluate bone turnover
Measurement of the following biomarkers in tumour tissue before and after the first AZD0424 administration: p-Src, MKI67 (Ki-67), p-PAX, p-CRKL, p-FAK.
Evaluate responses (stable disease (SD), partial response (PR) or complete response (CR)) in any of the patients as determined by Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Adrian Harris, Study Chair — Oxford University Hospitals NHS Trust
Locations (3):
- United Kingdom (3):
  - Belfast City Hospital, Belfast
  - Edinburgh Cancer Centre - Western General Hospital, Edinburgh
  - Oxford University Hospitals NHS Trust, Oxford

REFERENCES:
- [Derived] Woodcock VK, Clive S, Wilson RH, Coyle VM, Stratford MRL, Folkes LK, Eastell R, Barton C, Jones P, Kazmi-Stokes S, Turner H, Halford S, Harris AL, Middleton MR. A first-in-human phase I study to determine the maximum tolerated dose of the oral Src/ABL inhibitor AZD0424. Br J Cancer. 2018 Mar 20;118(6):770-776. doi: 10.1038/bjc.2017.484. Epub 2018 Feb 13. PMID 29438361